CLINICAL TRIAL: NCT00091676
Title: Randomized Trial of Patient-Specific Vaccination With Conjugated Follicular Lymphoma-Derived Idiotype (FNHLId1) With Local GM-CSF in First Complete Remission
Brief Title: Study of the BiovaxId Tumor Derived Idiotype Vaccine in Patients With Follicular Lymphoma
Acronym: BiovaxID
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biovest International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BV 301; NCT00001945 (obsolete NCT alias); NCT00019981 (obsolete NCT alias); NCT00096577 (obsolete NCT alias)
Record Dates: First submitted 2004-09-15; First posted 2004-09-17 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Non-Hodgkins Lymphoma
Keywords: follicular; lymphoma; Non-Hodgkins; idiotype; vaccine; indolent follicular Non-Hodgkins Lymphoma; tumor-derived; B-cell; cancer
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Neoplasms | interventions — keyhole-limpet hemocyanin; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ID-KLH + GM-CSF (Experimental)
  Interventions: Biological: FNHLId1
- KLH + GM-CSF (Active Comparator)
  Interventions: Biological: KLH + GM-CSF

INTERVENTIONS:
Biological: FNHLId1 — 5 monthly vaccinations over a 6 month time period consisting of 0.5 mg ID-KLH s.c. on day 1 and 100 mcg/m²/day GM-CSF s.c. on days 1-4
  Arms: ID-KLH + GM-CSF
Biological: KLH + GM-CSF — 5 monthly vaccinations at month 1, 2, 3, 4, and 6 consisting of 0.5 mg KLH s.c on day 1 and 100 mcg/m²/day GM-CSF s.c. on days 1-4
  Arms: KLH + GM-CSF

SUMMARY:
The primary objective of this Phase 3 study is to definitively confirm the safety and efficacy of BiovaxId, an autologous tumor derived immunoglobulin idiotype vaccine, as measured by a significant prolongation of the period of disease free survival when administered to patients with indolent follicular Non-Hodgkin's Lymphoma (NHL) during their first complete remission.

DETAILED DESCRIPTION:
Patients with Stage III-IV follicular lymphoma and tumor > 2cm (Stage II allowed if tumor > 5cm), previously untreated by other than local radiation, provide tumor material by tissue biopsy for production of a patient-specific Ig idiotype vaccine conjugated to the immunogenic protein KLH. After completing PACE or CHOP-R chemotherapy and achieving a complete remission, followed by a waiting period to reconstitute the immune system, patients who remain in remission randomized to the active treatment arm receive a series of 5 idiotype vaccinations accompanied by the immune stimulant GM-CSF. Patients randomized to the control arm receive a time-matched series of KLH injections also accompanied by GM-CSF. Patients are subsequently studied to observe their immune responses both to the non-specific immune stimulating agents and for the specific immune response to the vaccine. Patients are followed for a minimum of 4 years post-randomization or until relapse.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* Diagnosis of indolent follicular lymphoma(follicular small-cleaved cell, follicular mixed or follicular large cell with centrocytes) with surface IgM or IgG phenotype.
* Stage III-IV with lymph node > 2cm or Stage II with lymph node > 5 cm
* No prior chemotherapy other than local radiation (not greater than 2 sites)
* ECOG < 2
* Survival > 1 yr
* Serum creatinine < 1.5 mg/dl
* Bilirubin <1.5 mg/dl
* SGOT/SGPT < 3.5 ULN
* No HIV antibodies or HBV antigen
* Negative pregnancy screen (females)
* No unrelated neoplasm in the previous 10 years
* No evidence of primary or secondary CNS lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 629 (Estimated)
Dates: Start 2000-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To demonstrate prolongation of the period of Disease Free Survival (significant prolongation of the period of complete remission) in idiotype vaccine treated patients | until date of relapse

SECONDARY OUTCOMES:
To determine the ability of the idiotype vaccine to produce a molecular complete remission | once subject achieves molecular CR
To determine the impact of molecular disease free survival | until relapse
To assess the ability of the idiotype vaccine to generate an immunologic response against the NHL tumor | varies
To compare the overall survival of subjects randomized to receive either treatment | minimum 5 years from last subject randomized
To confirm the safety of 5 monthly injections of the vaccine with GM-CSF | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Carlos F Santos, PhD, Study Director — Biovest International; Stephen J Schuster, MD, Principal Investigator — University of Pennsylvania

REFERENCES:
- [Background] Hsu FJ, Caspar CB, Czerwinski D, Kwak LW, Liles TM, Syrengelas A, Taidi-Laskowski B, Levy R. Tumor-specific idiotype vaccines in the treatment of patients with B-cell lymphoma--long-term results of a clinical trial. Blood. 1997 May 1;89(9):3129-35. PMID 9129015
- [Background] Bendandi M, Gocke CD, Kobrin CB, Benko FA, Sternas LA, Pennington R, Watson TM, Reynolds CW, Gause BL, Duffey PL, Jaffe ES, Creekmore SP, Longo DL, Kwak LW. Complete molecular remissions induced by patient-specific vaccination plus granulocyte-monocyte colony-stimulating factor against lymphoma. Nat Med. 1999 Oct;5(10):1171-7. doi: 10.1038/13928. PMID 10502821
- [Background] Kwak LW, Campbell MJ, Czerwinski DK, Hart S, Miller RA, Levy R. Induction of immune responses in patients with B-cell lymphoma against the surface-immunoglobulin idiotype expressed by their tumors. N Engl J Med. 1992 Oct 22;327(17):1209-15. doi: 10.1056/NEJM199210223271705. PMID 1406793
- [Background] Dar MM, Kwak LW. Vaccination strategies for lymphomas. Curr Oncol Rep. 2003 Sep;5(5):380-6. doi: 10.1007/s11912-003-0022-x. PMID 12895388
- [Result] Schuster SJ, Neelapu SS, Gause BL, Janik JE, Muggia FM, Gockerman JP, Winter JN, Flowers CR, Nikcevich DA, Sotomayor EM, McGaughey DS, Jaffe ES, Chong EA, Reynolds CW, Berry DA, Santos CF, Popa MA, McCord AM, Kwak LW. Vaccination with patient-specific tumor-derived antigen in first remission improves disease-free survival in follicular lymphoma. J Clin Oncol. 2011 Jul 10;29(20):2787-94. doi: 10.1200/JCO.2010.33.3005. Epub 2011 May 31. PMID 21632504
- See also: Related Info — http://www.accentia.net/science_biovaxid.php
- See also: Related Info — http://www.biovest.com/